CLINICAL TRIAL: NCT00501085
Title: LAP-BAND AP Early Experience Trial (APEX)
Status: Completed | Type: Observational
Sponsor: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MedAff-LBAP201
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- LAP-BAND: Patients who receive the LAP-BAND AP Adjustable Gastric Banding System.
  Interventions: Device: LAP-BAND AP Adjustable Gastric Banding System

INTERVENTIONS:
Device: LAP-BAND AP Adjustable Gastric Banding System — Reduction of food intake due to creation of smaller stomach pouch.

SUMMARY:
The purpose of this study is to evaluate the LAP-BAND AP System in severely obese patients.

DETAILED DESCRIPTION:
The primary objective of this study was to collect additional information about the safety and effectiveness of the LAP-BAND AP System in a real-life clinical setting. Effectiveness was assessed through the collection of weight loss data, as well as other secondary effectiveness measurements. Safety was assessed by the incidence and severity of adverse events (AEs) related to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled to receive the LAP-BAND AP System
* Willingness to follow protocol requirements, including: the Informed Consent Form (ICF), Health Insurance Portability and Accountability Act (HIPAA) forms, follow-up schedule, completion of patient questionnaires.

Exclusion Criteria:

* Per the LAP-BAND AP System Directions For Use (DFU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 521 (Actual)
Dates: Start 2007-06; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apollo Endosurgery, Study Director — Apollo Endosurgery, Inc.
Locations (1):
- Apollo Endosurgery, Austin, Texas, United States

REFERENCES:
- [Derived] Ponce J, Taheri S, Lusco V, Cornell C, Ng-Mak DS, Shi R, Okerson T. Efficacy and safety of the adjustable gastric band - pooled interim analysis of the APEX and HERO studies at 48 weeks. Curr Med Res Opin. 2014 May;30(5):841-8. doi: 10.1185/03007995.2013.874992. Epub 2014 Jan 16. PMID 24328415
- [Derived] Fusco M, James S, Cornell C, Okerson T. Weight loss through adjustable gastric banding and improvement in daytime sleepiness: 2 year interim results of APEX study. Curr Med Res Opin. 2014 May;30(5):849-55. doi: 10.1185/03007995.2013.874991. Epub 2014 Jan 17. PMID 24328387
- [Derived] Shayani V, Voellinger D, Liu C, Cornell C, Okerson T. Safety and efficacy of the LAP-BAND AP(R) adjustable gastric band in the treatment of obesity: results at 2 years. Postgrad Med. 2012 Jul;124(4):181-8. doi: 10.3810/pgm.2012.07.2561. PMID 22913906

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 521 Subjects were enrolled (defined as signing the informed consent). 515 Subjects started treatment and underwent LAP-BAND implantation. 6 Subjects did not have the LAP-BAND implanted after enrolling and signing the informed consent.
Period: Overall Study
Arm/Group | LAP-BAND
Started | 515 (Number of participants who were treated with the LAP-BAND System.)
Completed | 83 (Number of participants completing 5 year follow-up visit.)
Not Completed | 432
Not completed — Lost to Follow-up | 195
Not completed — Withdrawal by Subject | 34
Not completed — Subject Decision | 1
Not completed — Revision Surgery | 7
Not completed — Explantation Surgery | 26
Not completed — Adverse Event | 4
Not completed — Non-Compliance | 24
Not completed — Study closed by sponsor | 109
Not completed — Other loss to follow-up | 32

BASELINE CHARACTERISTICS:
Population: The analysis population is defined as the number of subjects who underwent treatment with the LAP-BAND System.
Arm/Group | LAP-BAND
Number analyzed (Participants) | 515
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (10.89)
Age, Customized [Median (Full Range); unit: years]
  Median Age | 42.7 [18.5 to 70.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 422
  Male | 93
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0
  Black | 52
  Hispanic | 16
  Caucasian | 443
  Other (Native American or unspecified) | 3
  Missing | 1
Baseline Weight [Mean (Standard Deviation); unit: pounds (lbs)] | 273.9 (51.37)
Body Mass Index (BMI) at Baseline [Mean (Standard Deviation); unit: kg/m2] | 44.0 (6.25)
Baseline Excess Weight [Mean (Standard Deviation); unit: pounds (lbs)] — Excess weight is equal to subject weight minus ideal weight (ideal weight is based on having a BMI of 25)
  pounds (lbs) | 118.7 (42.46)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Excess Weight
Description: Subjects' Percent Excess Weight Loss (%EWL) from baseline over the 5 year period post LAP-BAND implantation was measured. Excess Weight = Baseline weight - Ideal weight, where ideal weight is based on a BMI of 25 kg/m2.
Time Frame: Baseline to 5 Years
Population: The analysis population is defined as all subjects treated with the LAP-BAND System.
Measure: Mean (Standard Deviation); unit: percentage of excess weight lost
Arm/Group | LAP-BAND
Number analyzed (Participants) | 515
percentage of excess weight lost
  %EWL from baseline 48 Weeks Post-Surgery (n=402) | -45.7 (21.26)
  %EWL from baseline 24 Months Post-Surgery (n=304) | -50.8 (26.70)
  %EWL from baseline 36 Months Post-Surgery (n=226) | -47.7 (30.21)
  %EWL from baseline 48 Months Post-Surgery (n=156) | -46.5 (27.23)
  %EWL from baseline 60 Months Post-Surgery (n=84) | -45.9 (26.80)

2. Secondary Outcome: Subject BMI From Baseline to 5 Years Post LAP-BAND Implantation
Description: Subjects' Body Mass Index (BMI) was recorded at each follow-up visit for the 5 years after LAP-BAND implantation.
Time Frame: Baseline to 5 years
Population: The analysis population is defined as all subjects treated with the LAP-BAND System.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | LAP-BAND
Number analyzed (Participants) | 515
kg/m2
  BMI at 48 Weeks Post-Surgery (n=402) | 35.9 (6.39)
  BMI at 24 Months Post-Surgery (n=304) | 34.8 (6.49)
  BMI at 36 Months Post-Surgery (n=226) | 35.2 (6.98)
  BMI at 48 Months Post-Surgery (n=156) | 35.1 (6.20)
  BMI at 60 Months Post-Surgery (n=84) | 35.2 (6.49)

3. Secondary Outcome: Subject Reported Satiety
Description: Subjects rated their level of hunger, satiety after meals, and desire to eat at all follow-up visits. Level of hunger was rated using a 6-point scale: 0 = not hungry at all to 5 = as hungry as I have ever felt. Satiety after meals was rated using a 6-point scale: 0 = not at all full to 5 = as full as I have ever felt. Desire to eat was rated using a 6-point scale: 0 = no desire at all to 5 = extremely strong desire.
Time Frame: Baseline to 5 Years
Population: The analysis population is defined as all subjects treated with the LAP-BAND System.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LAP-BAND
Number analyzed (Participants) | 515
units on a scale
  Level of Hunger at Baseline (n=487) | 2.1 (1.21)
  Level of Hunger at Month 60 (n=81) | 2.3 (1.18)
  Level of Fullness at Baseline (n=488) | 3.5 (1.19)
  Level of Fullness at Month 60 (n=81) | 3.3 (1.29)
  Level of Desire to Eat at Baseline (n=488) | 2.4 (1.19)
  Level of Desire to Eat at Month 60 (n=81) | 2.7 (1.19)

4. Secondary Outcome: Subject Reported Quality of Life
Description: Quality of Life was assessed using the Obesity and Weight-Loss Quality of Life Questionnaire (OWL-QOL-17). The OWL-QOL-17 is a survey of 17 questions, that rates quality of life on a scale of 0 (better) to 102 (lower).
Time Frame: Baseline to 5 Years
Population: The analysis population is defined as all subjects treated with the LAP-BAND System.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LAP-BAND
Number analyzed (Participants) | 515
units on a scale
  OWL-QOL-17 Score at Baseline (n=496) | 69.8 (19.98)
  OWL-QOL-17 Score at Month 60 (n=74) | 34.5 (24.50)

5. Secondary Outcome: Subject Reported Sleepiness (Epworth Sleepiness Scale)
Description: The Epworth Sleepiness Scale (ESS) is a questionnaire used to determine a subject's level of daytime sleepiness. Subjects rate his or her chances of dozing off in different situations, which are combined into a total ESS score that can vary between zero (low level of daytime sleepiness) and 24 (high level of daytime sleepiness).
Time Frame: Baseline to 5 years
Population: The analysis population is defined as all subjects treated with the LAP-BAND System.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LAP-BAND
Number analyzed (Participants) | 515
units on a scale
  Reported Sleepiness at Baseline (n=498) | 8.0 (4.23)
  Reported Sleepiness at Month 60 (n=79) | 5.0 (3.21)

ADVERSE EVENTS:
Time Frame: Adverse Event information was collected from the time of LAP-BAND implantation to 5 years (end of study).
Description: Adverse Event data was collected for the analysis population, defined as all subjects treated with the LAP-BAND System (N=515)
Arm/Group | LAP-BAND
Serious Adverse Events (participants affected / at risk) | 38/515
Other Adverse Events (participants affected / at risk) | 158/515
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAP-BAND (N=515)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Band erosion (Surgical and medical procedures) | 3 (3)
Band removal (Surgical and medical procedures) | 3 (3)
Band Slip (Surgical and medical procedures) | 15 (16)
Death (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Device Malfunction (General disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Fibrous Band Obstruction (General disorders) | 2 (2)
Gastric Erosion (Gastrointestinal disorders) | 1 (1)
Gastric Leak (Gastrointestinal disorders) | 1 (1)
Gastric Perforation (Gastrointestinal disorders) | 1 (1)
Gastric Prolapse (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Stomal Tumor (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Upset (Gastrointestinal disorders) | 1 (1)
Gastroesophageal Reflux Disease (GERD) (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Intra-abdominal Abscess (Gastrointestinal disorders) | 1 (1)
LapBand Port Revision (Surgical and medical procedures) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Sepsis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAP-BAND (N=515)
Acid Reflux (Gastrointestinal disorders) | 8 (9)
Band Slip (General disorders) | 4 (6)
Band too tight (General disorders) | 9 (19)
Cellulitis (Skin and subcutaneous tissue disorders) | 3 (3)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cholelithiasis (Renal and urinary disorders) | 5 (5)
Dilated Gastric Pouch (Gastrointestinal disorders) | 12 (22)
Dysphagia (Gastrointestinal disorders) | 37 (52)
Epigastric pain (Gastrointestinal disorders) | 4 (5)
Flipped Port (General disorders) | 6 (6)
Food Obstruction (Gastrointestinal disorders) | 4 (4)
Gastroesophageal Reflux Disease (GERD) (Gastrointestinal disorders) | 13 (17)
Heartburn (Gastrointestinal disorders) | 11 (13)
Increased Restriction (Gastrointestinal disorders) | 7 (7)
Pain at port site (General disorders) | 7 (7)
Port Tube Leaking (General disorders) | 3 (3)
Unable to tolerate solids/liquids (Gastrointestinal disorders) | 6 (9)
Vomiting/Nausea (Gastrointestinal disorders) | 42 (75)
Port Site Infection (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No